CLINICAL TRIAL: NCT02000024
Title: Assessing the Effectiveness of a Weight Watchers-based Lifestyle Intervention for the Primary Prevention of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: WW International Inc (Industry); Indiana Clinical and Translational Sciences Institute (Other); National Diabetes Education Program (Unknown)
Responsible Party: Principal Investigator, David Marrero, J.O Ritchey Professor of Medicine. Director, Diabetes Translational Research Center, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1109006877
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Prediabetes; Gestational Diabetes Mellitus; Obesity
MeSH Terms: conditions — Prediabetic State; Diabetes, Gestational; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle coaching (Experimental): The existing Weight Watchers lifestyle modification program including the online support tools.
  Interventions: Behavioral: Weight Watchers
- Lifestyle counseling (Active Comparator): Brief advice regarding risk factors and strategies to reduce them by lifestyle modification guided by National Diabetes Education Program (NDEP) materials.
  Interventions: Behavioral: Weight Watchers; Behavioral: National Diabetes Education Program

INTERVENTIONS:
Behavioral: Weight Watchers — The standard Weight Watchers program will serve as the base curriculum. Persons with increased risk for developing type 2 diabetes will be exposed to an initial "orientation session" designed to frame the rationale for participation in the program and to encourage attendance to a core series of sessions. This orientation session will reinforce the pre-diabetes status of participants and present the rationale for lifestyle modification as a means to reduce diabetes risk. In addition, this session will highlight the recommended sessions and topics that are needed to help reduce risk.
Behavioral: National Diabetes Education Program
  Arms: Lifestyle counseling

SUMMARY:
This study is a randomized pilot study to assess the applicability of the Weight Watchers model for lifestyle modification to the primary prevention of type 2 diabetes. The approach developed by Weight Watchers to achieve weight loss is based on similar nutritional principals and techniques used in the Diabetes Prevention Program (DPP) lifestyle intervention; monitoring food intake, exercising calorie control, setting modest weight loss goals and using physical activity.

DETAILED DESCRIPTION:
In the proposed study, the standard Weight Watchers program will serve as the base curriculum. Persons with increased risk for developing type 2 diabetes will be exposed to an initial "orientation session" designed to frame the rationale for participation in the program and to encourage attendance to a core series of sessions. This orientation session will reinforce the pre-diabetes status of participants and present the rationale for lifestyle modification as a means to reduce diabetes risk. In addition, this session will highlight the recommended sessions and topics that are needed to help reduce risk. In many respects it mirrors the curriculum content used in the DPP with regards to themes and specific topics. There are significant differences, however, between the two approaches that warrant investigation. Weight Watchers uses a point system to help users select appropriate foods. This system is less focused on fat gram control as a central theme than was the case with the DPP. More importantly, it uses an "open visit" system in which users get a core set of materials for home review that is then reviewed in facilitated group sessions. In this regard, the group session content is not configured as a sequential series of sessions delivered in a specific order, as was the case with the DPP. Moreover, participants can rejoin groups at any time that they choose. Weight Watchers also provides a sophisticated set of support materials online, using both phone apps (to help users track food consumption and "points" used) and a website program. The open attendance feature and the availability of online support should, in theory, facilitate long-term adherence.

ELIGIBILITY:
Inclusion Criteria:

* Persons age 18 and over
* Determination of BMI ≥ 24 kg/m2; persons of Asian Descent BMI ≥ 23 kg/m2
* Completion of the 7-item ADA Diabetes Risk Assessment and an ADA risk score ≥ 5
* Persons with a value of 100mg/dl or greater will confer eligibility from a single drop of whole blood obtained by finger stick to assess casual capillary blood glucose (CCBG) concentration using One-Touch Ultra handheld glucometer.
* Persons at high-risk for Impaired Glucose Tolerance (IGT), having an ADA Risk Score ≥5 and CCBG 110-199 mg/dl or an A1c ≥5.7%and < 6.5%.
* Women with a self-reported history of gestational diabetes with an A1c <6.5% and/or CCBG <199 mg/dl

Exclusion Criteria:

* Persons under the age of 18
* Persons with no evidence of pre-diabetes.
* Persons who are pregnant or planning to become pregnant.
* Person unable or unwilling to provide consent.
* Screening attendees who have a known condition that could alter glucose metabolism (e.g. pregnancy; known diabetes; antipsychotic or steroid medications; certain diseases or other conditions including Cushing's syndrome, acromegaly, pheochromocytoma, chronic pancreatitis, or HIV.)
* Heart attack, stroke or transient ischemic attack (TIA) in the past 6 months.
* Uncontrolled hypertension: systolic > 180 mm Hg or diastolic >105 mm Hg.
* Persons receiving treatment for cancer (excluding surgery alone) within the last 2 years(excluding skin cancer).
* Chest pain.
* Shortness of breath with minimal activity or at rest.
* Unexplained dizziness or fainting with physical activity (exercise).
* Chronic lung disease: Chronic Obstructive Pulmonary Disease (COPD) or asthma requiring home oxygen therapy (excluding sole use of a continuous positive airway pressure (CPAP) machine).
* Current use of anti-diabetes medications for the treatment of diagnosed diabetes
* Unable to communicate with research staff (including intervention staff).
* Unable to read written English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2011-12; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in weight | 6, 12, 19 and 24 months from baseline

SECONDARY OUTCOMES:
Changes in A1c | 6, 12, 19 and 24 months from baseline
Changes in systolic blood pressure | 6, 12, 19 and 24 months from baseline
Changes in total cholesterol | 6, 12, 19 and 24 months from baseline
Changes in HDL-cholesterol | 6, 12, 19 and 24 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: David G Marrero, Ph.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Marrero DG, Palmer KN, Phillips EO, Miller-Kovach K, Foster GD, Saha CK. Comparison of Commercial and Self-Initiated Weight Loss Programs in People With Prediabetes: A Randomized Control Trial. Am J Public Health. 2016 May;106(5):949-56. doi: 10.2105/AJPH.2015.303035. Epub 2016 Feb 18. PMID 26890171